CLINICAL TRIAL: NCT01083888
Title: ASP1517 Clinical Pharmacological Study Examination of Pharmacokinetics and Pharmacodynamics in Patients With Renal Anemia Undergoing Hemodialysis
Brief Title: ASP1517 Pharmacokinetics Study in Anemia Patients on Hemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1517-CL-0203
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Anemia; Hemodialysis; Renal Impairment
Keywords: FG-4592; ASP1517; Safety and tolerability; Plasma concentration; Pharmacokinetics
MeSH Terms: conditions — Anemia; Renal Insufficiency | interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 group (Experimental): Participants received a single oral dose of ASP1517 on Days 1 and 8
  Interventions: Drug: roxadustat

INTERVENTIONS:
Drug: roxadustat — oral
  Other Names: ASP1517

SUMMARY:
To assess the Pharmacokinetics and pharmacodynamics of single doses of ASP1517 in renal anemia patients on hemodialysis. Safety and tolerability will be also evaluated in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic renal failure patients receiving hemodialysis thrice weekly
* Body weight: >=40.0 and <80.0 kg
* Mean hemoglobin level >=10.0 and =<12.0 g/dL

Exclusion Criteria:

* Patients with severe inflammation or infection
* Patients who have a medical history of gastrointestinal surgery or enterectomy
* Patients who have uncontrolled hypertension
* Patients whose AST, ALT, total bilirubin, GGT exceed the ULN or those who have a medical history of serious liver diseases
* Patients who have a medical history of severe cardiac or cerebrovascular diseases
* Patients who have received blood transfusion or who have had a surgery (except surgery for a shunt) within 4 weeks
* Patients with a medical history of serious drug allergies
* Patients who may be pregnant or lactating, or who refuse to use required birth control during the study period

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-02-15 (Actual); Primary Completion 2010-06-07 (Actual); Study Completion 2010-06-07 (Actual)

PRIMARY OUTCOMES:
ASP1517 concentrations in plasma | For 96 hours after dosing

SECONDARY OUTCOMES:
ASP1517 concentrations in dialysate | For 6 hours after dosing
Plasma EPO level | Pre dosing and for 24 hours after dosing
Safety assessed by Adverse Event, vital signs standard 12-lead ECG or lab tests | For 96 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Chūbu, Japan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=353